CLINICAL TRIAL: NCT06554301
Title: A Study on the Efficacy and Safety of Empagliflozin in the Treatment of Pulmonary Arterial Hypertension
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: The Second Hospital of Shandong University (Other); The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCRCSZ-2023-015
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo in treatment pulmonary arterial hypertension (Placebo Comparator)
  Interventions: Drug: placebo in treatment pulmonary aerterial hypertension
- empagliflozin in treatment pulmonary arterial hypertension (Experimental)
  Interventions: Drug: empagliflozin in treatment pulmonary aerterial hypertension

INTERVENTIONS:
Drug: empagliflozin in treatment pulmonary aerterial hypertension — On the basis of background treatment, the experimental group was given 10 mg of empagliflozin tablets orally once a day for 12 weeks.
  Arms: empagliflozin in treatment pulmonary arterial hypertension
Drug: placebo in treatment pulmonary aerterial hypertension — On the basis of background treatment, the control group was given 10 mg of placebo tablets orally once a day for 12 weeks.
  Arms: placebo in treatment pulmonary arterial hypertension

SUMMARY:
The goal of this clinical trial is to learn if empagliflozin works to treat patients with pulmonary arterial hypertension. It will also learn about the safety of empagliflozin. The main questions it aims to answer are:

Based on standard treatment, does empagliflozin reduce pulmonary artery pressure and improve cardiac function in patients with pulmonary arterial hypertension? What medical problems do participants have when taking empagliflozin? Researchers will compare empagliflozin to a placebo (a look-alike substance that contains no drug) to see if empagliflozin works to treat patients with pulmonary arterial hypertension.

Participants will:

Take empagliflozin or a placebo every day for 12 weeks Visit the clinic once every 4 weeks for checkups and tests Keep a diary of their symptoms and the drug taking situation

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Sign the informed consent form.
3. Subjects who are willing and able to comply with the requirements of prescribed visits, treatment plans, laboratory examinations and other research procedures.
4. PAH with symptoms was initially diagnosed and belonged to one of the following subgroups:

   A. Idiopathic pulmonary hypertension (IPAH); B. hereditary pulmonary hypertension (HPAH); C drug or toxin-induced PAH, based on previous exposure to drugs, chemicals or toxins, such as fenfluramine derivatives, other appetite suppressants, toxic rapeseed oil or L- tryptophan.

   D. PAH is accompanied by:

   A) connective tissue disease B) Congenital systemic-pulmonary shunt (surgical correction must be performed at least one year before screening, and there is no or no clinically insignificant systemic-pulmonary shunt [1.0≤ lung-systemic blood flow ratio (QP/QS)≤1.5]), according to the opinion of the researcher.
5. Received right heart catheterization (RHC) at the time of screening or within 5 years before screening (if RHC is not performed, it will be performed during screening), which is consistent with the diagnosis of PAH and meets all the following criteria:

   A. mean pulmonary artery pressure (papm) > 20mmhg (at rest) B pulmonary arteriole wedge pressure (PAWP)≤15 mmHg (if reliable PAWP data cannot be obtained, left ventricular end diastolic pressure [LVEDP]≤15 mmHg).

   C pulmonary vascular resistance (PVR) > 2.00 wood units (> 160 dynes/sec/cm5).
6. There are symptoms of WHO/NYHA FC Grade II or III.
7. Stable PAH targeted background oral therapy. Subjects received endothelin receptor antagonist (ERA) and/or phosphodiesterase inhibitor type 5 (PDE5-I) or soluble guanylate cyclase (sGC) agonist. Stability was defined as no change in dose or regimen within 30 days before baseline and during the duration of the study.
8. 6-minute walking distance (6 MWD) ≥ 150m.
9. If the subject is taking concomitant drugs that can affect PAH (for example, calcium channel blockers, digoxin or L- arginine supplements), the dose must be kept stable for at least 30 days before the baseline visit and throughout the study.
10. If there is the possibility of pregnancy, both male and female subjects should agree to use a highly effective contraceptive method during the whole study period (from informed consent to the end of follow-up).

Exclusion Criteria:

* 1) Subjects shall not have the following three or more risk factors for left ventricular dysfunction: Body mass index (BMI)≥30 kg/m2 History of systemic hypertension

There is any of the following evidence to prove the history of major coronary artery disease:

A coronary angiographic evidence of a history of myocardial infarction or percutaneous coronary intervention or coronary artery disease (at least one coronary artery stenosis > 50%); B. Positive results of exercise provocation test and image evidence; C. previous coronary artery bypass surgery; D. stable angina pectoris; 2) Pulmonary function tests (PFTs) conducted within 180 days before or during the screening showed mild or above lung diseases. Subjects who meet any of the following criteria will be excluded: A. forced expiratory volume in the first second (FEV1)<60% (expected value); or B total lung volume (TLC) < 60% of the estimated value. 3) The evidence of thromboembolic disease is confirmed by lung ventilation/perfusion (V/Q) scanning or local standard diagnosis and treatment evaluation at the time of diagnosis or after diagnosis of PAH.

4) Severe chronic liver disease (i.e. Child-pugh grade C), portal hypertension, cirrhosis or complications of cirrhosis/portal hypertension (e.g., history of varicose bleeding, history of hepatic encephalopathy).

5) Confirm the active infection of hepatitis B virus (HBV) or hepatitis C virus (HCV).

6) Subjects whose alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level is more than or equal to 3 times the normal upper limit value (ULN) or whose total bilirubin is more than or equal to 2 times ULN at the time of screening.

7) Chronic renal insufficiency at screening, which is defined as serum creatinine > 2.5 mg/dL or requiring dialysis support.

8) Hemoglobin concentration < 9 g/dL during screening. 9) diabetes. 10) cardiac function grade IV (NYHA classification) 11) The subject has been treated with IV or SC prostacyclin pathway drugs (for example, epoprostol, triprostinil or iloprost) at any time before baseline (allowed to be used in pulmonary vasodilation test).

12) The subject has pulmonary vein occlusion disease. 13) Diagnosed and/or treated with malignant tumor within 5 years before screening, but excluding localized non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin, or radical resection of cervical carcinoma in situ.

14) At the time of screening, there was a history of alcohol or drug abuse within 6 months.

15) Start the exercise-based cardiopulmonary rehabilitation program within 90 days of the screening period and/or during the study period.

16) Participated in other interventional clinical studies within 30 days before screening. It is allowed to participate in registered or observational studies at the same time, as long as the subjects meet all other selection criteria and comply with all research process requirements.

17) Any reason (for example, any past or intermittent diseases) that the respondent thinks may increase the risk of participating in the study or may affect the study analysis and damage the study participation or collaboration, so that the subject cannot participate in the study.

18) Those who are known to be allergic to Engelgin or any auxiliary materials. 19) According to the researcher's judgment, life expectancy is less than 12 months.

20) Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
6-minute walking distance | From enrollment to the end of treatment at 12 weeks
  6-minute walking distance

SECONDARY OUTCOMES:
Clinical deterioration event | From enrollment to the end of treatment at 12 weeks
  Clinical deterioration event
Cardiac function index(NT-proBNP, WHO functional classification) | From enrollment to the end of treatment at 12 weeks
  Cardiac function index(NT-proBNP, WHO functional classification)
Hemodynamic index | From enrollment to the end of treatment at 12 weeks
  Hemodynamic index
Health-related quality of life (HRQoL) index | From enrollment to the end of treatment at 12 weeks
  Health-related quality of life (HRQoL) index
Cardiac magnetic resonance (CMR) | From enrollment to the end of treatment at 12 weeks
  Cardiac magnetic resonance (CMR)

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No